CLINICAL TRIAL: NCT06476509
Title: A Non-Randomized, Open-Label, Exploratory Mechanistic Validation (PoM) Clinical Trial of LV232 Capsule Assessing Serotonin Transporter Occupancy in the Healthy Adult Brain Using 11C-DASB Positron Emission Tomography (PET)
Brief Title: A Study to Assess Serotonin Transporter Occupancy of Healthy Adults Using 11C-DASB PET
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vigonvita Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LV232-03
Record Dates: First submitted 2024-06-18; First posted 2024-06-26 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LV232 (Experimental): A single oral dose of 40mg LV232 (5 mg/capsule, 8 capsules each time) ，administrated in fasting state, with 240 mL water to take A single oral dose of 60mg LV232 (5 mg/capsule, 12 capsules each time) ，administrated in fasting state, with 240 mL water to take A single oral dose of 20mg LV232 (5 mg/capsule, 4 capsules each time) ，administrated in fasting state, with 240 mL water to take
  Interventions: Drug: LV232 40mg; Drug: LV232 60mg; Drug: LV232 20mg
- Escitalopram (Active Comparator): A single oral dose of 20mg Escitalopram (10 mg/tablet, 2 tablets each time) , administrated with 240 mL water
  Interventions: Drug: Escitalopram 20 mg

INTERVENTIONS:
Drug: LV232 40mg — oral
  Other Names: LV232
  Arms: LV232
Drug: Escitalopram 20 mg — oral
  Other Names: Escitalopram
  Arms: Escitalopram
Drug: LV232 60mg — oral
  Other Names: LV232
  Arms: LV232
Drug: LV232 20mg — oral
  Other Names: LV232
  Arms: LV232

SUMMARY:
This study was a non-randomized, open-label clinical study to assess Serotonin transporter occupancy in the brain of healthy adults using 11C-DASB positron emission tomography (PET)

DETAILED DESCRIPTION:
This trial adopts a single-center, non-randomized, open-label design, with a planned enrollment of 16 healthy subjects. The LV232 capsule groups include 6 subjects in the 40 mg dose group, 4 subjects in the 60 mg dose group, and 4 subjects in the 20 mg dose group. Additionally, there are 2 subjects in the escitalopram oxalate tablet (positive control drug) group. Based on the results of the LV232 capsule study, the investigator and sponsor will jointly decide whether to proceed with the positive control group, using escitalopram oxalate tablets at a dose of 20 mg as the positive control drug.

ELIGIBILITY:
Inclusion Criteria:

* Those who voluntarily participate in and sign the informed consent form after understanding the purpose, content, process and possible risks of the trial;
* Male and female, aged 18 to 45 years at the time of signing the informed consent form;
* Body weight, male≥ 50.0 kg ,female≥ 45.0 kg ,and body mass index (BMI) 19.0 ~ 26.0 kg/m2 (including the boundary value) at screening;
* Able to maintain good communication with the investigator and comply with the lifestyle restrictions specified in the protocol and various requirements of the clinical trial (scheduled visits, laboratory tests and other trial procedures);
* Subjects and their partners must use effective non-pharmacological contraception (e.g., abstinence and condom with intravaginal spermicide) throughout the study and for 6 months after the end of the study, and must not donate sperm.

Exclusion Criteria:

* Known to have a history of allergy to any component of the investigational product or similar drugs, or allergic constitution (previous allergy to two or more foods or drugs);
* The subject with skin diseases or has a history of skin allergies;
* The subject has a current or past medical history judged by the investigator that may affect the clinical trial or dysfunction, including but not limited to a past or present central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders, etc. that require medical intervention or other diseases that are not suitable for clinical trials (such as a history of mental illness);
* Individuals with a history of epileptic seizures, or those with any (acute or chronic) history of mental illness and family history of mental illness, or those with a history of neurodegenerative diseases and family history of neurodegenerative diseases, such as Alzheimer's disease;
* Any surgical condition or condition that may significantly affect the absorption, distribution, metabolism and excretion of the drug, or may pose a hazard to the subjects participating in the trial; such as history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), urinary tract obstruction or dysuria, gastroenteritis, gastrointestinal ulcers, gastrointestinal bleeding, etc.;
* Abnormal vital signs (resting pulse rate<55 beats/minute or>100 beats/minute; Systolic blood pressure<90 mmHg or ≥ 140 mmHg; Diastolic blood pressure<60 mmHg or ≥ 90 mmHg), laboratory tests (blood routine , blood biochemistry, urine routine, thyroid Function), 12 electrocardiogram (ECG, male QTcF>450 ms，female QTcF>460 ms), MRI (magnetic resonance imaging) examination indicators, judged by the investigator as abnormal and clinically significant;
* Use of any prescription medication within 28 days prior to dosing; Use of any over-the-counter medications, including health products, within 7 days prior to dosing; Receipt of any contrast agent or radiopharmaceutical within 7 days prior to, or application of contrast agent within 24 hours after, administration of the trial drug;
* Contraindications to PET or MRI (magnetic resonance imaging) (including claustrophobia, alcohol allergy, cardiac pacemaker and nerve stimulator in the body, metal foreign body in the body or tracer component allergy, etc.);
* Any positive result of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), HIV antibody (HIV-Ab) and Toluidine red unheated serum test (Trust);
* Smoking habit (an average daily smoking of ≥ 5 cigarettes per day within 3 months before administration), drinking habit (an average weekly drinking of more than 14 standard units within 3 months before administration, 1 unit = 360 mL of beer or 45 mL of 40% spirits or 150 mL of wine). Subjects who cannot quit smoking or drinking in clinical trials.
* Individuals who have a history of drug dependence (including drug use) within one year prior to administration, or who have tested positive for urinary drug abuse screening (benzodiazepines, cocaine, methamphetamine, amphetamine, methadone, tetrahydrocannabinol acid, barbiturates, morphine, phencyclidine, tricyclic antidepressants);
* Those who have special requirements for food and cannot abide by the unified diet or have dysphagia;
* Consumption of xanthine-rich foods or beverages (e.g., tea, coffee, cola, or chocolate) or foods or beverages containing grapefruit and/or pomelo within 3 days before dosing;
* Significant occupational exposure to ionizing radiation (e.g., more than 50 millivolts per year) or exposure to radioactive substances or ionizing radiation for therapeutic or research purposes within the past year;
* Blood donation or blood loss ≥ 400 mL within 3 months before administration, or blood donation or blood loss ≥ 200 mL within one month;
* Those who have participated in other clinical trials within 3 months before administration (including drug and medical device clinical trials, the time is based on the last visit, except for those who have failed screening in other clinical trials and have not received any treatment);
* Pregnant, lactating women or male subjects whose spouses have a parenting plan within 3 months;
* Individuals who cannot tolerate intravenous administration ;
* Personnel directly related to this clinical trial;
* Patients with poor compliance or other problems who are not suitable for participating in this trial in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-01-19 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Serotonin Transporters occupancy | baseline and 3 hours after administration on Day 1
  Percentage of Serotonin Transporters Occupancy in Human Brain after oral LV232 capsule

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs). | Up to Day 7
  Incidence of treatment-emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng SHEN, MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center Ethics Committee, Shanghai, China

IPD SHARING:
Plan to Share IPD: No